CLINICAL TRIAL: NCT02759289
Title: Arsenic Exposure, Disordered Glucose Homeostasis and Atherosclerosis Protocol
Brief Title: Arsenic, Disordered Glucose Homeostasis and Atherosclerosis
Acronym: EMERALD-D
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 15-00725
Record Dates: First submitted 2016-04-27; First posted 2016-05-03 (Estimated); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Atherosclerosis; Type 2 Diabetes (T2D)
Keywords: Arsenic
MeSH Terms: conditions — Atherosclerosis; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A: Prediabetes glycohemoglobin test A1c 5.7-6.4%
- Group B: T2D glycohemoglobin test= A1c 6.5-7.9% without T2D medications
  T2D glycohemoglobin test=A1c ≥ 8.0% with/without T2D medications
- Group C: Control

SUMMARY:
Investigators will recruit 250 subjects; Group A will consist of 100 prediabetic patients with an A1c of 5.7%-6.4%. Group B will consist of 100 patients with uncontrolled T2D defined as either a) an A1c of 6.5%-7.9% without diabetes medications or b) an A1c ≥ 8.0% with or without diabetes medications. Group C will include 50 participants without T2D or known cardiovascular disease to serve as control comparisons.

DETAILED DESCRIPTION:
Patients with prediabetes have an elevated risk of cardiovascular disease (CVD). Cardiovascular disease (CVD) is also the leading cause of morbidity and mortality in patients with Type 2 Diabetes. There remains an unmet clinical need to identify modifiable risk factors for CVD in patients with disordered glucose homeostasis, including prediabetes and T2D. Exposure to inorganic arsenic and other environmental toxicants may be novel targets for CVD risk reduction for these patients. However, there have been no clinical studies of environmental exposures on vascular function and thrombotic risk among patients with prediabetes and growing understanding of environmental exposures as modifiable risk factors for CVD, and can have an impact by: (1) describing the role of environmental exposures for patients with or at risk for T2D; (2) identifying T2D patients at higher risk for the adverse biological effects of environmental exposures; and (3) informing health policies and treatment pathways to reduce the risk of these exposures.

Investigators will evaluate the association between inorganic arsenic exposure and measures of vascular function, estimate the association between inorganic arsenic exposure and measures of thrombotic risk and will explore the independent association between environmental exposures other than inorganic arsenic and measures of vascular function and thrombotic risk.

ELIGIBILITY:
Inclusion Criteria:

* No known cardiovascular, cerebrovascular or peripheral arterial disease
* Able and willing to provide written informed consent for the study

Exclusion Criteria:

* Unable to speak Spanish or English
* Active smoking (within the past year)
* Autoimmune, rheumatologic or inflammatory disease
* Known active cancer receiving treatment
* Pregnancy
* Anemia (hemoglobin < 9 mg/dl)
* Chronic kidney disease (CrCl < 30ml/min)
* Known Coronary Artery Disease (CAD; prior stents or CABG)
* Congestive Heart Failure
* Known Peripheral Arterial Disease (PAD; lower extremity revascularization surgery OR lower extremity stenting)
* Known prior stroke or transient ischemic attack (TIA) (mini-stroke or temporary/transient stroke)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Disordered Glucose Homeostasis
  * Group A: Prediabetes, A1c 5.7-6.4%
  * Group B: T2D A1c 6.5-7.9% without T2D medications T2D A1c ≥ 8% with/without T2D medications
  * Control patients (Group C): Normal glucose homeostasis
Sampling Method: Non-Probability Sample
Enrollment: 279 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Multiple linear regression to estimate the difference in brachial artery reactivity associated with a 1-Standard Deviation change in urinary arsenic | 6 Months, 12 Months
Change in platelet activity in response to arsenic exposure measured by Regression models | 6 Months, 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Newman, MPH, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States